CLINICAL TRIAL: NCT02409940
Title: A Randomized Trial to Elucidate Effect of Mesenchymal Stem Cells on Immune Modulation in Living Related Kidney Transplant Patients
Brief Title: To Elucidate the Effect of Mesenchymal Stem Cells on the T Cell Repertoire of the Kidney Transplant Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr. Aruna Rakha, DST Inspire Faculty, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IFA-LSBM-11
Record Dates: First submitted 2015-03-24; First posted 2015-04-07 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Renal Transplant Rejection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Autologus Mesenchymal Stem Cells (Experimental): This group would get two doses of mesenchymal stem cell (MSCs) infusion, one day pre transplant and 30 days post transplant. These MSCs would be derived from transplant recipient's bone marrow which are cultured in GMP compliant laboratories for 4-6 weeks.
  Interventions: Biological: Mesenchymal Stem Cells
- Allogeniec Mesenchymal Stem Cells (Active Comparator): This group would get two doses of mesenchymal stem cell (MSCs) infusion, one day pre transplant and 30 days post transplant. These MSCs would be derived from transplant donor's bone marrow which are cultured in GMP compliant laboratories for 4-6 weeks.
  Interventions: Biological: Mesenchymal Stem Cells
- Control without Mesenchymal Stem Cells (No Intervention): This group would get no stem cell infusion.

INTERVENTIONS:
Biological: Mesenchymal Stem Cells — These Mesenchymal stem cells are derived from bone marrow of either renal transplant patients or their donors depending upon the group of study.
  Other Names: Mesenchymal Stromal Cells
  Arms: Allogeniec Mesenchymal Stem Cells; Autologus Mesenchymal Stem Cells

SUMMARY:
Despite being a miracle of modern medicine, solid organ transplant recipients are always at risk of rejection, and remain dependent on lifelong immunosuppression. Currently used immunosuppressive drugs suppress the potential of immune system and interfere with the metabolism of medications. Cellular therapies currently being investigated for this purpose require the use of ablative radiotherapy. The investigators are using a less toxic strategy by harnessing the immunosuppressive potential of the MSCs in the Kidney Transplant (KTx) recipients and studying immunomodulation mediated by these cells in the KTx patients.

Hypothesis MSCs interfere with signalling of Immune cells like T cells, B cells and Dendritic cells which leads to improve graft survival of renal transplant patients.

Aim To investigate effect of MSCs on immune cell repertoire in a donor specific mediated response.

The investigators aim to collect peripheral blood from 30 patients (10 patients for autologous cell infusion and 10 for allogeneic (donor derived cell infusion) at various time intervals following MSC therapy. 10 patients serve as controls on standard dose of drugs but without MSC infusion. This peripheral blood would be utilized for isolation of mononuclear cells and performing various immune assays on these cells in a donor specific response.

DETAILED DESCRIPTION:
This is an open label type of study having 3 groups of patients: 1st group comprising of patients that would undergo allogeneic (donor-derived) mesenchymal stem cell infusion, 2nd group that would undergo autologous (patient-derived) mesenchymal stem cells and the third group (control group) without any stem cell infusion. All the three groups would have standard dose of Immunosuppressive drugs. Initially the investigators want to recruit 10 patients in each group and would increase the group size if the investigators get promising results on the follow up. The investigators plan to follow up the patients upto 1-2 years for immune based assays and then continue the follow up for atleast 5 years.

ELIGIBILITY:
Inclusion Criteria:

* All the renal transplant recipients participating in the trial should undergo primary kidney transplant.
* Donor should be living and related to the patient.
* Kidney transplant recipients and donor should be willing to give informed consent form.

Exclusion Criteria:

* There should be no prior sensitization to the patients.
* Patients should not be participating in any other study
* Patients should not be suffering from any autoimmune disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-09; Primary Completion 2016-09 (Actual); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Expansion of regulatory T cell compartment of the patients undergoing renal transplant and infused with mesenchymal stem cells as compared to the control patients. | 6 months
Normalization of serum creatinine levels of the patients undergoing renal transplant and infused with mesenchymal stem cells as compared to the control patients. | 6 months

SECONDARY OUTCOMES:
T cell proliferation changes in patients undergoing renal transplant and infused with mesenchymal stem cells as compared to the control patients. | 0day (one day before transpnatation), 30 days, 90days, 180 days, 1year, 2year post transplantation
Changes in regulatory T cells in patients undergoing renal transplant and infused with mesenchymal stem cells as compared to the control patients. | 0day (one day before transpnatation), 30 days, 90days, 180 days, 1year, 2year post transplantation
Changes in memory T cells in patients undergoing renal transplant and infused with mesenchymal stem cells as compared to the control patients. | 0day (one day before transpnatation), 30 days, 90days, 180 days, 1year, 2year post transplantation
Changes in B cells in patients undergoing renal transplant and infused with mesenchymal stem cells as compared to the control patients. | 0day (one day before transpnatation), 30 days, 90days, 180 days, 1year, 2year post transplantation
Changes in cytokine profile in patients undergoing renal transplant and infused with mesenchymal stem cells as compared to the control patients. | 0day (one day before transpnatation), 30 days, 90days, 180 days, 1year, 2year post transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Aruna Rakha, PhD., Principal Investigator — PGIMER, Chandigarh, India
Locations (1):
- Translational and Regenerative Medicine, Chandigarh, Chandigarh, India

REFERENCES:
- [Background] Mudrabettu C, Kumar V, Rakha A, Yadav AK, Ramachandran R, Kanwar DB, Nada R, Minz M, Sakhuja V, Marwaha N, Jha V. Safety and efficacy of autologous mesenchymal stromal cells transplantation in patients undergoing living donor kidney transplantation: a pilot study. Nephrology (Carlton). 2015 Jan;20(1):25-33. doi: 10.1111/nep.12338. PMID 25230334
- [Background] Rakha A, Todeschini M, Casiraghi F. Assessment of anti-donor T cell proliferation and cytotoxic T lymphocyte-mediated lympholysis in living donor kidney transplant patients. Methods Mol Biol. 2014;1213:355-64. doi: 10.1007/978-1-4939-1453-1_29. PMID 25173397